CLINICAL TRIAL: NCT07353190
Title: Comparison of the Effectiveness of TENS and TENS + NMES Treatment in Stroke Patients With Shoulder Pain: Prospective Randomized Controlled Study
Brief Title: Comparison of the Effectiveness of TENS and TENS + NMES Treatment in Stroke Patients With Shoulder Pain
Acronym: TENS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Park Bursa Hospital (Other)
Responsible Party: Principal Investigator, Sevinç Külekçioğlu, doctor lecturer, Medical Park Bursa Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-5/13
Record Dates: First submitted 2025-12-27; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Shoulder Disease; Hemiplegia; Hemiplegic Shoulder Pain
Keywords: stroke; shoulder pain; TENS; NMES
MeSH Terms: conditions — Stroke; Hemiplegia; Shoulder Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Electrical Nerve Stimulation (TENS) (Active Comparator): Participants in this group will receive Transcutaneous Electrical Nerve Stimulation (TENS) in addition to the standard stroke rehabilitation program. TENS application will be performed with appropriate electrode placement in the hemiplegic shoulder area for pain control. The intensity of application will be adjusted to a level that the participant can tolerate and will create a distinct sensory perception. Neuromuscular Electrical Stimulation (NMES) will not be applied in this group.
  Interventions: Procedure: TENS; Other: NMES
- Transcutaneous Electrical Nerve Stimulation (TENS) and Neuromuscular Electrical Stim (Active Comparator): Participants in this group will receive Transcutaneous Electrical Nerve Stimulation (TENS) in addition to the standard stroke rehabilitation program and Neuromuscular Electrical Stimulation (NMES) in addition to TENS. TENS application will be applied to the hemiplegic shoulder area for pain control. NMES application will be applied to target the paretic muscle groups involved in shoulder stabilization, aiming to achieve visible muscle contraction. It will be evaluated whether this combination provides additional clinical benefit in pain, shoulder function, and upper extremity use compared to TENS alone.
  Interventions: Procedure: TENS; Other: NMES

INTERVENTIONS:
Procedure: TENS — Transcutaneous Electrical Nerve Stimulation (TENS) will be applied to reduce hemiplegic shoulder pain. The stimulation will be delivered to the hemiplegic shoulder region using appropriate electrode placement. TENS parameters, including frequency, pulse duration, and treatment duration, will be set according to standard clinical practice. Stimulation intensity will be adjusted to produce a clear but comfortable sensory perception without causing discomfort. TENS will be administered in addition to the standard stroke rehabilitation program.
Other: NMES — Neuromuscular Electrical Stimulation (NMES) will be applied in addition to TENS to activate paretic muscle groups involved in shoulder stabilization. NMES will be delivered to target muscles in order to elicit visible muscle contractions. Stimulation parameters, including frequency, pulse duration, contraction-relaxation cycles, and total treatment time, will be determined in accordance with standard clinical practice and adjusted based on participant safety and tolerance. NMES will be provided as an adjunct to both TENS and the standard stroke rehabilitation program.

SUMMARY:
In this study, the effects of Transcutaneous Electrical Nerve Stimulation (TENS) and Neuromuscular Electrical Stimulation (TENS + NMES) applied in addition to TENS on pain, shoulder joint range of motion and upper extremity functions will be comparatively evaluated in stroke patients with hemiplegic shoulder pain. In this direction, in the study; The effectiveness of both treatment approaches on the severity of hemiplegic shoulder pain, their contribution to shoulder functionality and daily living activities will be examined; It will be investigated whether NMES application added to TENS provides an additional clinical benefit compared to TENS.

DETAILED DESCRIPTION:
Hemiplegic shoulder pain that develops after stroke is a common complication that negatively affects upper extremity functions, shoulder joint range of motion (ROM) and daily living activities. Muscle weakness accompanying the pain, loss of activation of the shoulder girdle muscles, subluxation, spasticity and limitation of movement; It may delay the recovery process by reducing rehabilitation participation. While Transcutaneous Electrical Nerve Stimulation (TENS), one of the electrophysical agents, is a widely used method in pain modulation, Neuromuscular Electrical Stimulation (NMES) has the potential to increase paretic muscle activation, support shoulder stabilization and improve functional gains. However, there is limited evidence as to whether NMES added to TENS provides additional clinical benefit in hemiplegic shoulder pain.The aim of this randomized controlled clinical study was to compare TENS and TENS + NMES applications in stroke patients with hemiplegic shoulder pain; To evaluate the effects on (i) pain intensity, (ii) shoulder joint range of motion, (iii) upper extremity functions and (iv) daily living activities. The main hypothesis of the study is that NMES added to TENS will provide a greater reduction in pain and a more significant improvement in shoulder function/upper extremity use compared to TENS alone.

Study Design

This study is a prospective, parallel group, randomized controlled clinical trial to be conducted in stroke patients with hemiplegic shoulder pain. Participants will be divided into two branches:

TENS Group: TENS will be applied in addition to the standard rehabilitation program.

TENS + NMES Group: TENS will be applied in addition to standard rehabilitation; Additionally, NMES will be applied in addition to TENS.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 and over
* Patients with a history of clinically and radiologically confirmed ischemic or hemorrhagic stroke
* Hemiplegic shoulder pain in the affected shoulder
* Shoulder pain severity VAS/NRS ≥ 2
* At least 2 weeks and at most 1 year have passed since the onset of stroke
* Have a level of cognitive and communicative competence that will not hinder the application of clinical evaluations and scales
* Must have signed the Informed Volunteer Consent Form to participate in the study.
* Must have a general medical condition to participate in a conventional rehabilitation program

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 4 weeks
  Hemiplegic Shoulder Pain Severity; The severity of shoulder pain on the hemiplegic side will be evaluated using the visual analogue scale VAS. Participants will rate their pain level from 0 (no pain) to 10 (the worst pain imaginable). Pain assessment will be performed at rest and/or during shoulder movement.

IPD SHARING:
Plan to Share IPD: No